CLINICAL TRIAL: NCT01725477
Title: Laparoscopic Tubal Patency Assessment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pourmatroud, Elham, M.D. (Individual)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: Methylen blue; Methylen blue in laparoscopy (Registry Identifier: PourmatroudE)
Record Dates: First submitted 2012-10-25; First posted 2012-11-12 (Estimated); Last update posted 2017-04-11 (Actual); Status verified 2017-04

CONDITIONS: Methylene Blue; Laparoscopy; Tubal Patency
MeSH Terms: interventions — Saline Solution; Coloring Agents; Methylene Blue

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dye& normal saline/ 20ml methylene blue +50 ml normal saline (Experimental): first arm:20 ml methylene blue washing with50 ml normal saline
  Interventions: Drug: methylen blue &normal saline; Drug: methylene blue; Drug: metheylne blue with normal saline
- injection of 20ml metheylen blue (Active Comparator): 20 ml methylene blue injected without washing
  Interventions: Drug: methylene blue

INTERVENTIONS:
Drug: methylen blue &normal saline — Washing after dye injection
  Other Names: DYE; Methylene BLUE
  Arms: Dye& normal saline/ 20ml methylene blue +50 ml normal saline
Drug: methylene blue
Drug: metheylne blue with normal saline
  Arms: Dye& normal saline/ 20ml methylene blue +50 ml normal saline

SUMMARY:
1. Methylene blue in laparoscopy use for tubal patency assessment
2. Methylene blue could have negative effect on sperm motility, oocyte granulosa cell and fertility.
3. tubal washing after Methylene blue administration could be effective in pregnancy rate after operation.

DETAILED DESCRIPTION:
women with unexplained infertility and without any problem during laparoscopy and hysteroscopy entered in the study.After randomization in one group after dye test,washing with normal saline was done until all of visible Methylene blue removed.In second group washing with normal saline did not done. pregnancy rate until three months after operation was followed without any intervention.

ELIGIBILITY:
Inclusion Criteria:

* women with unexplained infertility

Exclusion Criteria:

* any intervention during operation like ovarian drilling or septum resection

Ages: 20 Years to 38 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2012-09; Primary Completion 2014-02-14 (Actual); Study Completion 2015-03-09 (Actual)

PRIMARY OUTCOMES:
Pregnancy rate | up to 12 weeks

SECONDARY OUTCOMES:
complications rate in two group | Up to 12 weeks

OTHER OUTCOMES:
Abortion rate | Up to 12 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Ahvaz Jundishapur university of medical science, Ahvāz, Iran

REFERENCES:
- [Result] Galili Y, Ben-Abraham R, Rabau M, Klausner J, Kluger Y. Reduction of surgery-induced peritoneal adhesions by methylene blue. Am J Surg. 1998 Jan;175(1):30-2. doi: 10.1016/s0002-9610(97)00232-8. PMID 9445235